CLINICAL TRIAL: NCT01228929
Title: Non-invasive Ocular Surface Measurements Before and After Interventions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, James V. Aquavella, MD, Principal Investigator, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 32315
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Dry Eye Syndrome; Healthy
Keywords: Dry Eye; Non-invasive instruments; MGD; Environment; Thermal Imaging
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal (Experimental): Subjects with no clinical diagnosis or symptoms of dry eye.
  Interventions: Other: Environmental Chamber Condition Change Intervention
- Aqueous Deficiency Dry Eye (ADDE) (Experimental): Subjects with low tear volume measured by Schirmer's test less than 10 mm.
  Interventions: Other: Environmental Chamber Condition Change Intervention
- Meibomian Gland Dysfunction (MGD) (Experimental): Subjects having mild to moderate Meibomian Gland Dysfunction by slit lamp evaluation.
  Interventions: Other: Environmental Chamber Condition Change Intervention

INTERVENTIONS:
Other: Environmental Chamber Condition Change Intervention — For condition change studies, the chamber will operate between 65 and 85 degrees F and 25% and 80% RH with air flow turned off or set to a maximum of 3-4 m/s. For this type of study, we will have the subject acclimate to a set of environmental conditions (approximately 20-30 minutes) and take a set of measurements. Then we will change the conditions (rate of change is 3 degrees F/hour and 3% RH/hour), have the subject acclimate to these conditions (later on the same day or on another day) and take another set of measurements. The expected study length is approximately two hours for a single visit. Subjects may be asked to return for additional visits to accommodate a variety of chamber conditions (temp, humidity, airflow) within the prescribed limits above.

SUMMARY:
Objectively evaluate the ocular surface (pre-corneal tear film) of individuals prior to and after an intervention (such as a dry eye treatment, environmental change, artificial tear use, or contact lens wear) in a controlled-environmental chamber, over time using non-contact instruments.

DETAILED DESCRIPTION:
Most studies will set the environmental conditions (temperature, humidity, airflow) to mimic typical office and home environments (68 to 72F and 20 to 50%). For condition change studies, the chamber will operate between 65 and 85F and 25% and 80% RH with air flow turned off or set to a maximum of 3-4 m/s. For this type of study we will have the subject acclimate to a set of environmental conditions (approximately 20 minutes) and take a set of measurements. Then we will change the conditions (rate of change is 3F/hour and 3% RH/hour), have the subject acclimate to these conditions (later on the same day or on another day) and take another set of measurements. The expected study length is approximately two hours for a single visit.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with dry eye diagnoses (aqueous deficient dry eye [ADDE], and/or evaporative dry eye), dry eye symptoms (as associated with Sjogren's Syndrome diagnosis), refractive surgery, contact lens use, and exposure to dry work environments are appropriate to correlate clinical tests, subjective responses and objective measurements of current ocular surface status and to study clinically-recommended or patient-directed dry eye treatments such as taking dietary supplements, wearing moisture-retaining goggles, performing lid massage, or using over the counter eye drops or artificial tears.
* Individuals who do not currently have dry eye symptoms but who may be at risk for dry eye diagnosis, and those who have dry eye symptoms but no clinical dry eye diagnosis, are of interest to correlate clinical tests, subjective responses and objective measurements of current ocular surface status and, if symptoms appear or worsen, to correlate the data with the effect of environmental condition changes, such as increasing the humidity or reducing air flow, on the ocular surface.
* Individuals who have undergone ocular surgery are at increased risk for dry eye. While some subjects who have had ocular surgery may never develop dry eye symptoms because they have an adequate reserve of tear production, others may develop symptoms as a result of the disruption of the ocular surface, including the anatomy and nerves. Subjects who have had surgery or procedures and are no longer being provided with direct post-operative care may participate in the study. Routine follow-up post- operative care does not disqualify subjects from participation. Subjects who are receiving post-operative care must obtain approval of their clinician to participate in the study.
* Individuals who have eye conditions that affect the shape or condition of the cornea, such as individuals with keratoconus.
* Experienced contact lens wearers are appropriate for studies that use their own lenses (soft, rigid gas permeable [RGP], hard [PMMA]) or the same type of lens within the FDA approved modality (daily, continuous or extended wear) and replacement cycle (for example, daily, one week, one month, etc.) as described in the lens package insert and/or prescribed by their eye care provider to investigate ocular surface data before, during and after lens use.
* Normal individuals, those without a dry eye diagnosis, without dry eye symptoms or those who do not wear contacts to act as controls for the focus areas in the studies.

Exclusion Criteria:

Individuals with eye or medical condition(s) that contraindicate performing screening or measurements will not be eligible for this study. Specific examples include:

* Individuals will not be dilated if an exam and/or medical history indicted they have a narrow anterior chamber angle, glaucoma, or other contraindications to dilation (like arterio-sclerotic cerebrovascular disease).
* Individuals with the following will not participate in contact lens studies: presence of ocular or systemic allergies or disease (infection), clinically significant (grade 3 or 4) corneal edema, corneal vascularization, or any other abnormalities of the cornea, tarsal abnormalities or bulbar injection or use of medication that might interfere with contact lens wear.
* Individuals will not participate in any aspect of the study if: they are pregnant or become pregnant or are lactating, have an infectious disease (e.g. hepatitis, tuberculosis) or have an immuno-suppressive disease (e.g. HIV).
* Individuals with known sensitivity to dyes or to numbing drops will not be screened using these agents.
* Individuals who wear dental braces cannot be involved in the measurements in which a dental impression/bite bar is required. The impression material will stick to the braces. Individuals with very sensitive teeth or loose dentures may have difficulty making the dental impression.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James V Aquavella, MD, Principal Investigator — University of Rochester
Locations (1):
- Flaum Eye Institute at the University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal: Subjects with no clinical diagnosis or symptoms of dry eye. Each participant completed 3 environmental conditions. Nominal is 75 degrees F and 40% relative humidity. Low humidity is 20% relative humidity and 75 degrees F. High temperature is 85 degrees F and 40% relative humidity.
- Aqueous Deficiency Dry Eye (ADDE): Subjects with low tear volume measured by Schirmer's test less than 10 mm. Each participant completed 3 environmental conditions. Nominal is 75 degrees F and 40% relative humidity. Low humidity is 20% relative humidity and 75 degrees F. High temperature is 85 degrees F and 40% relative humidity.
- Meibomian Gland Dysfunction (MGD): Subjects having mild to moderate Meibomian Gland Dysfunction by slit lamp evaluation. Each participant completed 3 environmental conditions. Nominal is 75 degrees F and 40% relative humidity. Low humidity is 20% relative humidity and 75 degrees F. High temperature is 85 degrees F and 40% relative humidity.
Period: Nominal Condition
Arm/Group | Normal | Aqueous Deficiency Dry Eye (ADDE) | Meibomian Gland Dysfunction (MGD)
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0
Period: Low Humidity Condition
Arm/Group | Normal | Aqueous Deficiency Dry Eye (ADDE) | Meibomian Gland Dysfunction (MGD)
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0
Period: High Temperature Condition
Arm/Group | Normal | Aqueous Deficiency Dry Eye (ADDE) | Meibomian Gland Dysfunction (MGD)
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal | Aqueous Deficiency Dry Eye (ADDE) | Meibomian Gland Dysfunction (MGD) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 18
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 9
  Male | 2 | 4 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Ocular Surface Temperature (OST)
Description: Objectively evaluate the ocular surface temperature prior to and after 30 minutes of acclimation to three different environmental conditions in a controlled-environmental chamber using thermal imaging. 10 eyes were analyzed for each group.
Time Frame: baseline and 30 minutes
Measure: Mean (Standard Deviation); unit: degree celsius
Units Other Than Participants: eyes
Arm/Group | Normal | Aqueous Deficiency Dry Eye (ADDE) | Meibomian Gland Dysfunction (MGD)
Number analyzed (Participants) | 6 | 6 | 6
Number analyzed (eyes) | 10 | 10 | 10
degree celsius
  Nominal | 0.047 (0.03) | 0.020 (0.03) | 0.127 (0.04)
  Low humidity | 0.015 (0.02) | 0.062 (0.02) | 0.013 (0.03)
  High temperature | -0.060 (0.02) | 0.064 (0.02) | -0.011 (0.02)

ADVERSE EVENTS:
Arm/Group | Normal | Aqueous Deficiency Dry Eye (ADDE) | Meibomian Gland Dysfunction (MGD)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes